CLINICAL TRIAL: NCT03368209
Title: Noninvasive Glucose Measurements - Database and Calibration Compilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to recruit sufficient subjects
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-07
Record Dates: First submitted 2017-11-22; First posted 2017-12-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes
Keywords: Non-invasive glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Open, non-randomized comparison study between device and blood references with diabetic patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OUH protocol (Experimental): The protocol constituted two outpatient visits in the clinic within one week. Each visit had a duration of approximately 2,5 hours. Prior to study, optical screenings were conducted:
  * Optical Coherence Tomography (OCT)
  * Optical screening on measuring site with WM3.4.
  Subjects were measured by the following scheme: ABL measurement, two optical measurements on WM3.4 #1 followed by two optical measurements on WM3.4 #2.
  Interventions: Device: WM3.4
- Home 1 protocol (Experimental): Optical screening (OCT and device) was conducted at baseline visit in the Department of Endocrinology M at Odense University Hospital.
  WM3.4 was subsequently delivered to subject's home and the subject measured 30 days in a 60 days period of time. HemoCue was used for reference.
  Interventions: Device: WM3.4
- Home 2 protocol (Experimental): Optical screening (OCT and device) was conducted at baseline visit in the Department of Endocrinology M at Odense University Hospital.
  WM3.4 was subsequently delivered to subject's home and the subject measured 30 days in a 60 days period of time. HemoCue and CGM/FGM was used for reference.
  Interventions: Device: WM3.4

INTERVENTIONS:
Device: WM3.4 — Investigational Medical Device collecting spectral raman data from tissue.

SUMMARY:
This study collected spectral raman data from diabetic patients. Data was paired with validated capillary references as well as CGM/FGM readings. Data was used to develop models for glucose prediction.

DETAILED DESCRIPTION:
This trial constitutes three subprotocols: "The OUH protocol", "The Home 1 protocol" and "The Home 2 protocol" The investigation was initiated to collect spectral raman data paired with validated blood references. In the OUH protocol, capillary blood was analysed by ABL 800 Flex blood gas analyzer by Radiometer. In the Home 1 protocol, references were obtained by the finger pricking procedure from HemoCue (Radiometer). In the Home 2 protocol, HemoCue measurements were conducted along with continuous monitoring using Dexcom G4/G5 device (Dexcom) or FreeStyle Libre (Abbott) The data was collected from diabetic patients and Optical Coherence Tomography (OCT) readings were obtained from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with and without diabetes including pregnant women

Exclusion Criteria:

* Subject under 18 years of age
* Subjects not able to understand provided information
* Subjects without measuring sites
* Subjects with rash or wound on measuring sites
* Subjects with stained fingers, such a oil or nicotine
* Subjects not capable of holding arm/hand steadily on probe
* Subjects with thrombosis in arm/hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-07 (Actual)

PRIMARY OUTCOMES:
Calibration models for device predictive purposes | 6 months
  Spectral raman data paired with validated references used to develop predictive algorithms with glucose prediction capablities. The preformance was validated using the consensus error grid.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, Principal Investigator — Odense University Hospital, Dpt. of Endocrinology M
Locations (1):
- Department of Endocrinology M, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No